CLINICAL TRIAL: NCT02098694
Title: Physiotherapy-led Outpatient Clinic for Patients With Spondyloarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: Helse Møre og Romsdal HF (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013/1520 (REK)
Record Dates: First submitted 2014-03-25; First posted 2014-03-28 (Estimated); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Spondylarthritis; Spondylitis, Ankylosing; Spondylarthropathies; Sacroiliitis; Arthritis, Psoriatic
Keywords: Physiotherapy; Outpatient clinic
MeSH Terms: conditions — Spondylarthritis; Spondylitis, Ankylosing; Spondylarthropathies; Sacroiliitis; Arthritis, Psoriatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physiotherapy follow-up (Experimental): Consultation at Physiotherapy-led Outpatient Clinic every 4 month.
  Interventions: Other: Physiotherapy follow-up
- Usual care (No Intervention): Consultation every 4 months, twice a year by rheumatologist as usual, once a year by nurse.

INTERVENTIONS:
Other: Physiotherapy follow-up — Physiotherapy consultation every 4 months containing assessment of the spine and its mobility, including axial joints, assessment of the patients activity profile.
  Instruction in home-exercises and recommendations for optimization of activity profile. Information regarding the disease and the importance of physical activity and exercise.
  Arms: Physiotherapy follow-up

SUMMARY:
The purpose of this study is to determine whether patients with spondyloarthritis are more satisfied with a physiotherapy-led outpatient clinic than usual care and whether there is a difference between patients in a physiotherapy-led outpatient clinic and those in usual care regarding disease activity, function and mobility.

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis spondyloarthritis, ankylosing spondylitis, spondylarthropathy, juvenile ankylosing spondylitis, psoriatic arthritis with affection of the spine
* age between 18 and 45 (born 1969 - 1996)

Exclusion Criteria:

* also diagnosed with potentially functionally impairing neuromuscular, neurological or muscular disorders
* insufficient Norwegian language skills
* cognitive impairment
* no sign of inflammation or bone erosions in the sacroiliac joints or in the spine on imaging

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Leeds Patient Satisfaction Questionnaire (LSQ) | 8 months

SECONDARY OUTCOMES:
Bath Ankylosing Spondylitis Metrology Index (BASMI) | 8 months
Bath Ankylosing Spondylitis Functional Index (BASFI) | 8 months
Ankylosing Spondylitis Disease Activity Score (ASDAS) | 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Ann-Katrin Stensdotter, PhD, Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- Department of Rheumatology, Ålesund hospital, Ålesund, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Holoyen PK, Stensdotter AK. Patients with spondyloarthritis are equally satisfied with follow-up by physiotherapist and rheumatologist. Musculoskeletal Care. 2018 Sep;16(3):388-397. doi: 10.1002/msc.1241. Epub 2018 Mar 24. PMID 29573538